CLINICAL TRIAL: NCT00825890
Title: The High Cup/Disc Ratio in Children
Status: Completed | Type: Observational
Sponsor: Kim's Eye Hospital (Other)
Responsible Party: Principal Investigator, Ungsoo Kim, Professor, Kim's Eye Hospital
Other Study IDs: USK-1
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma
Keywords: high cup disc ratio; glaucoma suspect
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To investigate of high cup/disc ratio in children.

DETAILED DESCRIPTION:
ophthalmologic examination

1. cycloplegic refraction
2. axial length and anterior chamber depth
3. intraocular pressure

B. optic nerve head and retinal nerve fiber layer

1. disc photography
2. Heidelberg Retina Tomograph

ELIGIBILITY:
Inclusion Criteria:

* high cup/disc ratio more than 0.5
* age : five to twelve

Exclusion Criteria:

* previous surgery (except strabismus surgery) previous glaucomatous medication history poor cooperated children.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: high cup disc ratio in children
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ungsoo S Kim, M.D., Principal Investigator — Kim's Eye Hospital, University of Konyang
Locations (1):
- Kim's Eye Hospital, Seoul, Seoul, South Korea